CLINICAL TRIAL: NCT00350584
Title: Evaluation of Two Telehealth Interventions Targeting Post-Trauma Stress in Combat Veterans: Comparing Mindfulness and Psychoeducation
Brief Title: Evaluation of Telehealth Interventions for Post-Trauma Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Boston Healthcare System (U.S. Federal Agency)
Collaborators: Samueli Institute for Information Biology (Other)
Responsible Party: Barbara L. Niles, Ph.D., Principal Investigator, VA Boston Healthcare System, National Center for PTSD
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Telehealth for PTSD Symptoms; SIIB 1 EA-0000043
Record Dates: First submitted 2006-07-10; First posted 2006-07-11 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2009-01

CONDITIONS: Post Traumatic Stress Disorders
Keywords: Mindfulness; Psychoeducation; Telehealth Intervention
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness Telehealth for PTSD (Experimental): Participants receive two in-person sessions and 6 sessions over the phone. Participants are introduced to mindfulness concepts. CDs with guided meditation exercises are given to participants and they are asked to practice between sessions.
  Interventions: Behavioral: Mindfulness Telehealth Intervention
- Psychoeducation Telehealth for PTSD (Active Comparator): Participants receive two in-person sessions and six telehealth sessions with education about symptoms of PTSD and coping strategies. In addition, participants are asked to read short homework assignments and think about them during the week; these are discussed in weekly sessions.
  Interventions: Behavioral: Psychoeducation Telehealth Intervention

INTERVENTIONS:
Behavioral: Mindfulness Telehealth Intervention — Two in-person sessions and six telephone sessions with a therapist. Focus is on learning mindfulness skills.
  Arms: Mindfulness Telehealth for PTSD
Behavioral: Psychoeducation Telehealth Intervention — Two in-person sessions and six telephone sessions with a therapist. Focus is on education about PTSD.
  Arms: Psychoeducation Telehealth for PTSD

SUMMARY:
Posttraumatic Stress Disorder (PTSD) is very prevalent within the veteran population and is associated with decreased quality of life and an increased risk of developing other psychiatric and physical illnesses. The overarching objective of the proposed study is to evaluate the effectiveness of two telehealth treatment conditions in promoting healing within a population of veterans with full or partial PTSD. In particular, we are targeting newly returned veterans from the Iraq and Afghanistan conflicts. Specifically, we are comparing the relative efficacy of an alternative therapeutic approach, a Mindfulness based treatment, with a Psychoeducation treatment in reducing symptoms of PTSD and more generalized psychiatric symptoms, while increasing quality of life. Of note, both treatment conditions will consist of two in-person sessions and six brief weekly telephone calls. Participants will be 58 veterans (29 per condition) recruited from the VA Boston Healthcare System. Assessment will occur before and after the delivery of the intervention. We hypothesize that while both treatments will result in improved outcomes, the Mindfulness intervention will promote more healing than the Psychoeducation intervention. Results from this project will help further our understanding of the role of mindfulness in treating PTSD, particularly in those veterans who are returning from deployment.

DETAILED DESCRIPTION:
Aim: To evaluate the relative feasibility and healing efficacy of two eight-week telehealth interventions for individuals with combat-related PTSD: (1) Mindfulness and (2) Psychoeducation.

Objectives:

1. The first short-term objective is to determine whether two eight-week telehealth interventions are:

   1. feasible to conduct in a population of veterans with symptoms of combat-related PTSD;
   2. effective at promoting healing specific to combat survivors as evidenced by reductions in symptoms of PTSD;
   3. effective at promoting more generalized healing in combat veterans as evidenced by reductions in symptoms that are often co-morbid with PTSD (e.g., depression, anxiety, and substance abuse problem severity); and
   4. effective at promoting healing beyond a symptom level in combat veterans as evidenced by increases in quality of life after the interventions.
2. The second short-term objective of this study is to determine whether a Mindfulness intervention will be more effective at promoting healing than a Psychoeducation intervention. This comparison will be made on the levels of specific PTSD symptoms, more general co-morbid symptoms, and global quality of life.
3. The long-term objectives of this line of research are to identify mechanisms of action in a Mindfulness Telehealth Intervention that allow healing and promote increased quality of life in individuals with PTSD.
4. An additional long-term objective of this project is to contribute to the development of efficacious wellness interventions that can promote healing after combat exposure in veterans returning from current military conflicts (e.g. Iraq and Afghanistan).

Hypotheses:

1. It is hypothesized that both eight-week telehealth interventions (Mindfulness and Psychoeducation) will be feasible in a population of veterans with symptoms of combat-related PTSD. Specifically, satisfaction and compliance with the interventions is predicted to be high.
2. It is hypothesized that both eight-week telehealth interventions (Mindfulness and Psychoeducation) will be effective at promoting healing and reducing symptoms of PTSD. Specifically, it is predicted that levels of PTSD measured post-intervention will be lower than levels measured pre-intervention.
3. It is hypothesized that both eight-week telehealth interventions (Mindfulness and Psychoeducation) will be effective at promoting healing and reducing symptoms co-morbid with PTSD. Specifically, it is predicted that levels of depression, anxiety, and substance abuse problem severity measured post-intervention will be lower than levels measured pre-intervention.
4. It is hypothesized that both eight-week telehealth interventions (Mindfulness and Psychoeducation) will be effective at improving quality of life. Specifically, it is predicted that levels of quality of life measured post-intervention will be higher than levels measured pre-intervention.
5. Although it is hypothesized that both eight-week interventions will be effective at healing for veterans with PTSD symptoms, the holistic Mindfulness intervention is hypothesized to be more effective at promoting healing and reducing symptoms of PTSD and co-morbid disorders and improving quality of life than the Psychoeducation intervention. Specifically, it is predicted that levels of PTSD, depression, anxiety, and substance abuse problem severity will be lower post-intervention and quality of life will be higher for those individuals in the Mindfulness condition than for those in the Psychoeducation condition.

ELIGIBILITY:
Inclusion Criteria:

* documented United States military service in war or peacekeeping theater
* a current diagnosis of PTSD or partial PTSD
* access to a telephone

Exclusion Criteria:

* veteran's mental status precludes completion of the assessment procedures (e.g., severe organicity or active psychosis)
* the veteran's regimen of psychiatric medication has not been stable over the past two months (if applicable)
* the veteran has symptoms consistent with a diagnosis of alcohol or drug dependence within the past three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-02; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS) | pre and post intervention
  Gold standard instrument to assess symptoms of PTSD. Administered by a clinician.

SECONDARY OUTCOMES:
PTSD Checklist | pre and post intervention
  Self-report instrument to assess symptoms of PTSD.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara L Niles, Ph.D., Principal Investigator — VA Boston Healthcare System; Amy K Silberbogen, Ph.D., Principal Investigator — VA Boston Healthcare System
Locations (1):
- VA Boston Healthcare System, Boston, Massachusetts, United States